CLINICAL TRIAL: NCT03692000
Title: Digitally Supporting Lifestyle Changes in Men With Prostate Cancer - Part 2: User-driven Design and Development of a Digital Tool to Support Healthy Lifestyle in Men With Prostate Cancer Based on an Ethnographic Study of the Target Group
Brief Title: Designing a Digital Tool to Support Healthy Lifestyle in Men With Prostate Cancer
Acronym: Emil2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Danish Cancer Society (Other)
Collaborators: University of Copenhagen (Other); TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Dorthe Furstrand, Principal Investigator, Danish Cancer Society
Other Study IDs: DCS-53232017-2
Record Dates: First submitted 2018-09-29; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Health Literacy; Computer Literacy; Prostate Cancer
Keywords: eHealth Literacy; Health Literacy; Computer Literacy; Software Design; Healthy Lifestyle; Health Behavior
MeSH Terms: conditions — Prostatic Neoplasms; Health Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men with a history of prostate cancer: Men with a history of prostate cancer invited to participate in design-workshops , interviews or usabilitytesting.

SUMMARY:
The emil project aims to design, develop, implement and evaluate a digital service to support a healthy lifestyle among men with prostate cancer.

In this second study, men with a history of prostate cancer are invited to participate in the scoping and design of a digital platform, through three iterations of workshops and individual interviews, which includes prototyping and other ideation processes.

Finally, the men with a history of prostate cancer will be involved in the usability testing of the design, to ensure a platform fit for use by the intended users.

DETAILED DESCRIPTION:
In this user-driven study, the methods will be workshops, interviews, usability testing and a concluding proof of concept testing.

Workshops constitutes the bigger part of the user-driven design and ideation in this project. In workshops a group of people will generate a synergy that opens up for new ideas in a framed setting. The workshop format uses methods such as affinity diagrams; innovation jams; and ideation guided through artefacts such as Lego or paper cuts, with the researcher as the facilitator. After analysing the outcome of each design iteration, the findings will be incorporated into the design and focus the planning of the succeeding workshops in an iterative process.

The usability of the design will be tested in between workshops in interviews. The test will be performed by think aloud testing with the current prototype, recording for data collection and researchers in the room to observe, facilitate and probe for reflection.

For a more elaborate usability testing to conclude the design phase, a proof of concept will be performed. In this living lab scenario, the tool will be used at home by end-users in the intended way. Issues with technical functionality, user interphase, data management and workflow will surface and can be corrected during the proof of concept, thus consolidating the service before the feasibility study. Data collection from this part of the study will be by ongoing dialogue with participants, by e-mail and telephone.

To provide the broadest possible foundation for recruitment in terms of diversity in lifestyle and socioeconomic status, invitation to the study is done by mail directly to a randomly chosen group of men with prostate cancer.

All iterations will be based on the results of the previous. The first iteration is based on the ethnographic input from the first study.

All participants in study 2 will be met with a baseline questionnaire to evaluate digital readiness and e-health literacy and adjust participant configuration to ensure diversity. The questionnaire include self-reported educational level, health issues, treatments, diet, physical activity level and other lifestyle factors as well as eHLQ as part of the READHY questionnaire toolkit. The 13 dimensions of READHY comes from heiQ, HLQ and eHLQ, and work as a multidimensional validated robust psychometric instrument evaluation and can be used in combination to describe user's health technology readiness level and degree of enablement.

Each activity of the user-driven design process will be documented in a report, that will serve as the data foundation for a scientific publication.

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study will be men with prostate cancer, included in the Danish Cancer Registry under the IDC-10 code DC61 in the years 2014 or 2015.
* All participant will have registered residence in eastern Denmark, either in the Capital Region or in Region Zealand.

Exclusion Criteria:

* Men with known non-localized prostate cancer at the time of diagnosis. Non-localised cancer will be defined by use of the TNM classification in the Danish Cancer Registry as proposed by Outzen et al [17]: Tis1-4,x and N1-3 and M0,1,x or Tis 1-4,x and N0,x and M1.
* Participants will be excused from participation if they do not have sufficient written and spoken Danish language skills for participation in the activities involved in the studies. The researcher will assess whether the participants have sufficient cognitive functions to participate in the study, including be able to contribute to design workshops or report on everyday living. The researcher can also judge from an ethical perspective that the participant, for reasons not stated in the protocol, should be excused from participation in the study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Danish population
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Digital health service intervention design | 5 months. Each iteration of workshops and interviews evaluated to inform the next. Data evaluation points each month.
  The primary outcome is a design product which supports men in their everyday life to have a healthy lifestyle through digital means.
  A process of 3 iterations of workshops and individual interviews produces data in the form of notes, sketches, pictures, recordings and prototype-products. By iterative analysis and confirmation and ideation in the following iteration, the primary outcome of this process is the design of a digital health service intervention to support men with prostate cancer in a healthy lifestyle.

SECONDARY OUTCOMES:
Identification of digital capabilities and attitude of men with prostate cancer, in their everyday life | 5 months.
  Analysis of digital capabilities and attitude of the participants, from notes, sketches, pictures, recordings and prototype-products of the workshops and interviews.
Wireframe and mockup | 3 months
  Wireframe and mockup of the intervention, illustrated in the mockup-design tool Mockingbot (mockingbot.com).
Beta-test | 2-5 weeks
  Analysis of feedback from a beta-testing of the intervention design. Data collected via e-mail and telephone dialogue with the testers.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Tjønneland, MD PhD DMSc, Study Director — Danish Cancer Society Research Center; Lars Kayser, MD PhD, Study Chair — University of Copenhagen, Dept. of Public Health
Locations (1):
- Danish Cancer Society Research Center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
It is a priority to protect the privacy of participant according to research ethics guidelines and GDPR. Participant data will only be shared in anonymized form and only in the extend demanded by a journal.